CLINICAL TRIAL: NCT04440631
Title: Investigation of the Microbiome of Patients Receiving Antibiotic Therapy for Orthopedic Device-related Infection
Brief Title: Gut Microbiome of Patients Undergoing Antibiotic Therapy for Orthopedic Device-related Infection
Acronym: IMPAT-ODRI
Status: Completed | Type: Observational
Sponsor: AO Research Institute Davos (Other)
Responsible Party: Sponsor
Other Study IDs: Microbiome
Record Dates: First submitted 2020-05-14; First posted 2020-06-19 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Fractures, Bone; Infection, Bacterial; Joint Infection; Bone Infection
Keywords: Gut Microbiome; Joint Infection; Bone Infection; Antibiotic Therapy
MeSH Terms: conditions — Fractures, Bone; Bacterial Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Antibiotic therapy including rifampicin
  Interventions: Other: no intervention, observational only
- Non-rifampicin antibiotic therapy
  Interventions: Other: no intervention, observational only
- Control group (healthy volunteers)
  Interventions: Other: no intervention, observational only

INTERVENTIONS:
Other: no intervention, observational only — no intervention, observational only

SUMMARY:
The microbiome of 80 orthopedic-device related infection (ODRI) patients treated with antibiotics and 10 healthy controls will be investigated. Samples (blood, stool, saliva, skin-swab) are collected 4x within 6 months. Composition and diversity of the microbiome will be assessed by 16sRNA sequencing, skins swabs are screened for rifampicin-resistant staphylococci onto Mannitol-salt-agar plates supplemented with rifampicin, inflammation markers and antibodies in blood and saliva are monitored to track changes in the immune response. For further analysis patients are assigned to one of two groups: 1) antibiotic therapy including rifampicin and 2) non-rifampicin antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* The patient is planned to undergo revision surgery due to suspected bone or joint infection.
* The patient is at least 18 years old

Exclusion Criteria:

* The patient took antibiotics in the previous six weeks of recruitment (a single dose/"shot" of antibiotics during this period is not considered).
* The patient suffers from gut-associated morbidities such as Morbus Crohn or colitis ulcerosa.
* The patient suffers from psychiatric disorders/cognitive impairment affecting understanding.
* The patient is unable to give consent and follow procedures and/or has insufficient knowledge of the project language.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The project population will include patients suffering from an ODRI (orthopedic device-related infection). This includes any patient with a bone infection with a current or previous involvement of an implant. The majority of patients are expected to be prosthetic joint infection (PJI) and fracture-related infection (FRI) patients, although also patients with spinal implantation with an infection, or patients who have had an implant removed yet develop an osteomyelitis will also be included.
  These patients all have a deep bone implant infection and will receive antibiotic therapy, including at least two weeks IV therapy and at least 4 weeks of oral rifampicin. The investigators expect the distribution of patients getting rifampicin or non-rifampicin to be approximately 50/50 overall and anticipate PJI patients will be older, receive more concomitant medications and have underlying co-morbidities than patients with an FRI.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Composition of the the gut microbiota following two weeks of intravenous antibiotic therapy | Two weeks
  The gut microbiota will be characterized by means of 16s rRNA sequencing. The gut microbiota composition following two weeks of intravenous (iv) antibiotic treatment will be compared to baseline samples of the patients.
Composition of the gut microbiota following four weeks of oral antibiotic therapy | Six weeks (including two weeks iv and four weeks of oral antibiotic therapy)
  The gut microbiota will be characterized by means of 16s rRNA sequencing. The gut microbiota composition following four weeks of oral antibiotic treatment will be compared to baseline samples of the patients.
Composition of the gut microbiota 24 weeks after antibiotic therapy start | 24 weeks
  The gut microbiota will be characterized by means of 16s rRNA sequencing. The gut microbiota composition 24 weeks after antibiotic therapy start, including an at least 6-week antibiotic free period, will be compared to baseline samples of the patients.

SECONDARY OUTCOMES:
Monitoring Rifampicin resistant S. aureus on the skin following two weeks of iv antibiotic therapy | Two weeks
  Skin and nose swabs will be plated on (rifampicin supplemented ) Mannitol-Salt-Agar plates and colonies will be compared to baseline samples of the patients.
Monitoring Rifampicin resistant S. aureus on the skin following four weeks of oral antibiotic therapy | Six weeks (including two weeks iv and four weeks of oral antibiotic therapy)
  Skin and nose swabs will be plated on (rifampicin supplemented ) Mannitol-Salt-Agar plates and colonies will be compared to baseline samples of the patients.
Monitoring Rifampicin resistant S. aureus on the skin 24 weeks after antibiotic therapy start | 24 weeks
  Skin and nose swabs will be plated on (rifampicin supplemented ) Mannitol-Salt-Agar plates and colonies will be compared to baseline samples of the patients.

OTHER OUTCOMES:
Level of systemic Inflammation following two weeks of iv antibiotic therapy | Two weeks
  Inflammatory cytokines in the blood will be measured and compared to baseline samples of the patients.
Level of systemic Inflammation following four weeks of oral antibiotic therapy | Six weeks (including two weeks iv and four weeks of oral antibiotic therapy)
  Inflammatory cytokines in the blood will be measured and compared to baseline samples of the patients.
Level of systemic Inflammation 24 weeks after antibiotic therapy start | 24 weeks
  Inflammatory cytokines in the blood will be measured and compared to baseline samples of the patients.
Monitoring mucosal immune response following two weeks of iv antibiotic therapy | Two weeks
  IgA levels will measured in saliva of the patients and compared to baseline samples of the patients.
Monitoring mucosal immune response following four weeks of oral antibiotic therapy | Six weeks (including two weeks iv and four weeks of oral antibiotic therapy)
  IgA levels will measured in saliva of the patients and compared to baseline samples of the patients.
Monitoring mucosal immune response 24 weeks after antibiotic therapy start | 24 weeks
  IgA levels will measured in saliva of the patients and compared to baseline samples of the patients.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Schulthess Klinik Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided